CLINICAL TRIAL: NCT02492269
Title: Stress Response and Neurodevelopmental Outcome After Cardiac Surgery Utilizing CPB in Children: A Prospective, Double Blinded and Randomized Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aymen N Naguib (Other)
Responsible Party: Sponsor-Investigator, Aymen N Naguib, Director of Pediatric Cardiothoracic Anesthesia, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB13-00088
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Results first posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine in addition to 15 µg/kg of fentanyl
  Interventions: Drug: Dexmedetomidine
- Placebo (Placebo Comparator): Normal saline as a placebo in addition to 15 µg/kg of fentanyl
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Placebo
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
The overall goal of this project is to determine the role of anesthetic management in children undergoing cardiac surgery utilizing CPB in the setting of fast tracking and early extubation. An ideal anesthetic technique would ensure abolishing or diminishing stress response as would be evident by the stress markers levels and the level of two cerebral injury biomarkers (S 100 B and NSE). This should translate to better immediate postoperative outcome and hopefully improve both the short and the long term neurodevelopmental outcome in these children. The project is prospective, randomized and blinded study. The first and second aim of the study should be conducted over 2 year period. Our long term aim will be concluded when these children reach the school age.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following diagnosis:

  1. ASD
  2. VSD
  3. AVSD
  4. TOF
  5. Biventricular repair with left to right shunt.

Exclusion Criteria:

* Patients with the diagnosis of AVSD and pulmonary hypertension
* Patients less than 1 year and require any of the following repairs:

  1. HLHS
  2. Aortic arch reconstruction
  3. Arterial switch
  4. TOF with pulmonary atresia

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine: Dexmedetomidine in addition to 15 µg/kg of fentanyl
  Dexmedetomidine
- Placebo: Normal saline as a placebo in addition to 15 µg/kg of fentanyl
  Placebo
Period: Overall Study
Arm/Group | Dexmedetomidine | Placebo
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Placebo | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 16 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 6 (2) | 6 (2) | 6 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
Diagnosis [Count of Participants; unit: Participants]
  Ventricular Septal Defect | 7 | 5 | 12
  Tetralogy of Fallot | 6 | 9 | 15
  Atrioventricular septal defect | 6 | 2 | 8
Weight [Mean (Standard Deviation); unit: kilograms] | 6 (1) | 7 (1) | 6.6 (1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cytokine Levels
Description: Cytokine levels in plasma samples will be measured at induction of anesthesia (baseline), after sternotomy, after initiation of CPB, at the conclusion of surgery (separation from CPB and administration of protamine and prior to skin closure) and at 24 hours post-operatively.
Time Frame: From baseline to 24 hrs post-op
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 14 | 16
picograms per milliliter
  Baseline TNF-alpha | 4.38 (1.63) | 4.2 (2.55)
  Post-sternotomy TNF-alpha | 3.98 (1.58) | 3.85 (2.37)
  Post-bypass TNF-alpha | 2.88 (1.14) | 2.72 (1.76)
  End of surgery TNF-alpha | 3.12 (1.94) | 2.96 (1.7)
  24 hr. post-op TNF-alph | 2.68 (1.25) | 3.30 (2.43)
  Baseline IL-6 | 0.57 (0.71) | 0.96 (1.59)
  Post-sternotomy IL-6 | 0.61 (0.53) | 0.99 (1.29)
  Post-bypass IL-6 | 0.87 (0.59) | 1.19 (1.3)
  End of surgery IL-6 | 11.95 (21.71) | 11.32 (14.73)
  24 hr. post-op IL-6 | 30.2 (17.04) | 41.93 (74.34)
  Baseline IL-8 | 6.55 (5.02) | 7.28 (5.61)
  Post-sternotomy IL-8 | 6.8 (4.68) | 8.46 (6.03)
  Post-bypass IL-8 | 7.04 (5.26) | 8.35 (5.94)
  End of surgery IL-8 | 28.83 (28.97) | 34.37 (32.76)
  24 hr. post-op IL-8 | 20.86 (16.76) | 32.52 (29.81)
  Baseline IL-10 | 0.27 (0.62) | 0.9 (0.65)
  Post-sternotomy IL-10 | 0.87 (0.46) | 1.26 (0.89)
  Post-bypass IL-10 | 1.05 (1.02) | 1.24 (0.88)
  End of surgery IL-10 | 44.41 (48.95) | 78.27 (54.11)
  24 hr. post-op IL-10 | 1.37 (0.51) | 1.62 (1.03)

2. Primary Outcome: Change in Hormone Levels
Description: ACTH, cortisol, epinephrine, & norepinephrine will be measured at induction of anesthesia (baseline), after sternotomy, after initiation of CPB, at the conclusion of surgery (separation from CPB and administration of protamine and prior to skin closure) and at 24 hours post-operatively.
Time Frame: From baseline to 24 hrs post-op
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 14 | 16
picograms per milliliter
  Baseline ACTH | 150.10 (119.78) | 139.48 (96.11)
  Post-sternotomy ACTH | 105.63 (141.15) | 94.2 (93.8)
  Post-bypass ACTH | 108.09 (114.86) | 199.34 (160.34)
  End of surgery ACTH | 186.69 (170.06) | 201.49 (171.01)
  24 hr. post-op ACTH | 18.21 (9.8) | 26.78 (19.19)
  Baseline Cortisol | 448.27 (187.73) | 293.92 (138.53)
  Post-sternotomy Cortisol | 449.71 (144.4) | 316.58 (264.12)
  Post-bypass Cortisol | 314.42 (81.66) | 298.64 (217.82)
  End of surgery Cortisol | 553.88 (220.52) | 474.66 (256.16)
  24 hr. post-op Cortisol | 344.83 (344.79) | 357.3 (475.88)
  Baseline Epinephrine | 108.26 (98.2) | 112.13 (145.52)
  Post-sternotomy Epinephrine | 250.1 (261.97) | 379.68 (344.15)
  Post-bypass Epinephrine | 830.45 (757.89) | 830.73 (488.22)
  End of surgery Epinephrine | 203.73 (103.58) | 423.06 (406.03)
  24 hr. post-op Epinephrine | 172.05 (235.48) | 154.05 (176.39)
  Baseline Norepinephrine | 492.58 (475.2) | 696.5 (568.89)
  Post-sternotomy Norepinephrine | 545.88 (656.81) | 891.86 (966.44)
  Post-bypass Norepinephrine | 499.37 (428.34) | 1145.05 (1281.1)
  End of surgery Norepinephrine | 229.32 (207.5) | 477.66 (745.6)
  24 hr. post-op Norepinephrine | 913.12 (950.97) | 1320.9 (2263.32)

3. Primary Outcome: Change in Bayley Cognitive Composite Scores
Description: Children will have a baseline neurodevelopmental Bayley score during the preoperative period. These children will be retested prior to discharge from the hospital, at their post-op cardiology visit (usually 1-3 months post-op), six month and one year postoperatively to evaluate neurodevelopment progress.
  Mean score of 100 (SD=15) at the 50th percentile signifies mid-average functioning, scores below 85 (1 SD below the mean), at the 16th percentile, indicate mild impairment of being 'at risk' of developmental delay.
  Score below 70 (2 SD below the mean), at the second percentile, indicate moderate to severe impairment.
Time Frame: From baseline to 1 year post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 14 | 16
score on a scale
  Baseline | 102.14 (11.04) | 95 (16.12)
  Prior to discharge | 102.14 (13.26) | 88.33 (17.49)
  1-3 month post-op | 102.86 (14.9) | 96.82 (17.07)
  6 months post-op | 98.57 (7.95) | 97.27 (16.49)
  1 yr. post-op | 94.64 (12.0) | 94.09 (12.0)

4. Secondary Outcome: Change in Bayley Language Composite Scores
Description: as for outcome 3
Time Frame: From baseline to 1 year post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 14 | 16
score on a scale
  Baseline | 98.14 (13.95) | 86.81 (14.45)
  Prior to discharge | 91.14 (20.0) | 77.6 (12.26)
  1-3 month post-op | 92.5 (13.35) | 92.36 (14.43)
  6 months post-op | 86 (11.81) | 91.36 (8.98)
  1 yr. post-op | 93.08 (13.1) | 91.2 (18.64)

5. Secondary Outcome: Change in Bayley Motor Composite Scores
Description: Children will have a baseline neurodevelopmental Bayley score during the preoperative period. These children will be retested at their post-op cardiology visit (usually 1-3 months post-op), six month and one year postoperatively to evaluate neurodevelopment progress.
  Mean score of 100 (SD=15) at the 50th percentile signifies mid-average functioning, scores below 85 (1 SD below the mean), at the 16th percentile, indicate mild impairment of being 'at risk' of developmental delay.
  Score below 70 (2 SD below the mean), at the second percentile, indicate moderate to severe impairment.
Time Frame: From baseline to 1 year post-op
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dexmedetomidine | Placebo
Number analyzed (Participants) | 14 | 16
score on a scale
  Baseline | 95.14 (15.02) | 84.2 (15.89)
  1-3 month post-op | 92.07 (13.9) | 84.27 (16.84)
  6 months post-op | 92 (13.98) | 87.18 (10.66)
  1 yr. post-op | 91.69 (10.62) | 87.5 (17.37)

ADVERSE EVENTS:
Time Frame: 48 hours after surgery
Arm/Group | Dexmedetomidine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT02492269/Prot_SAP_000.pdf